CLINICAL TRIAL: NCT03601143
Title: Liquid Biopsy-based Detection of Resistance to Targeted Therapy in Prostate Cancer Patients
Acronym: PEARL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: HE 7386/1-1
Record Dates: First submitted 2018-07-02; First posted 2018-07-26 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-04

CONDITIONS: Castration-resistant Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood samples prior to a new line of AR-targeted therapy — Blood will be drawn at baseline prior to a new line of AR-targeted therapy.

SUMMARY:
This study will prospectively compare liquid-biopsy based methods for prediction of resistance under androgen-receptor signaling inhibitors. The main goal is to determine the optimal method to determine androgen-receptor variant 7 (AR-V7) status. In addition, the investigators will explore novel other, AR-V7 independent mechanisms of resistance and their predictive value for proper treatment. These are based on further AR splice variants, and on neuroendocrine differentiation of prostate cancer cells.

DETAILED DESCRIPTION:
Androgen receptor signaling inhibitors (ARSi) have become available in the past years for the treatment of patients with metastatic castration-resistant prostate cancer (mCRPC) and have significantly improved their survival. Despite this improvement, initial or emerging resistance to ARSi poses a major challenge in the treatment of these patients. There is therefore an urgent medical need for early detection of treatment resistance.

Liquid biopsies - blood samples containing circulating tumor cells (CTCs) and nucleic acids from the tumor - can provide information about such resistance. The investigators of this study and others have shown that liquid biopsies can be used to detect the messenger RNA (mRNA) of AR-V7, a splice variant of the androgen receptor (AR) that is insensitive to ARSi, in whole blood, and that high levels of AR-V7 mRNA in mCRPC patients are predictive to non-response to ARSi. Several liquid biopsy approaches involving different blood compartments such as CTCs, exosomes, and whole blood have been used so far to detect AR-V7. However, it is unclear which liquid biopsy approach or which combination of approaches is best to predict resistance under ARSi therapy in the clinical setting. In addition, current approaches explain only about half of resistant cases, suggesting that there are important non-AR-V7-mediated causes of resistance.

In this study, the investigators aim at determining the optimal liquid biopsy approach to detect AR-V7 and exploring novel ones for best possible prediction of resistance to ARSi. To this end, the investigators will systematically explore relevant blood compartments in a prospective cohort of mCRPC patients, quantify AR-V7 mRNA levels in each compartment, and determine the diagnostic value of compartment-specific AR-V7 mRNA levels for predicting response to subsequent ARSi therapy. The investigators will further explore the clinical relevance of AR-V7 protein subcellular localization in CTCs for prediction of ARSi resistance. In addition, novel other, AR-V7 independent mechanisms of resistance and their predictive value for proper treatment will be explored. These are based on further AR splice variants, and on neuroendocrine differentiation of prostate cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma
* Castrate serum testosterone <50ng/ml or <1.7nmol/l under continued androgen-deprivation therapy or surgical castration
* Progressive disease at study entry in accordance with Prostate Cancer Working Group 3 criteria (PCWG3):

  * Biochemical progression: Three consecutive rises in PSA at least one week apart resulting in two 50% increases over the nadir, and a PSA >1.0 ng/ml as minimal starting value, or
  * Radiologic progression: either two or more new bone lesions on bone scan or a new soft tissue lesion using RECIST (Response evaluation criteria in solid tumors).
* Metastatic disease confirmed on computed tomography (CT) or bone scan
* Planned treatment with ARSi (androgen-receptor signaling receptors)
* Written informed consent of the patient

Exclusion Criteria:

* Persons who are in a dependency or employment relationship with the investigator or sponsor
* Planned additional concurrent anticancer therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: metastatic castration-resistant prostate cancer patients planned for a new line of therapy with androgen-receptor signaling inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prostate-specific antigen (PSA) decline >=50% | 24 months
  The optimal liquid biopsy-based test method to predict PSA response under AR-targeted therapy will be determined.

SECONDARY OUTCOMES:
Clinical progression-free survival | 24 months
  The optimal liquid biopsy-based test method to predict clinical progression-free survival under AR-targeted therapy will be determined.
Overall survival | 36 months
  The optimal liquid biopsy-based test method to predict overall survival under AR-targeted therapy will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias M Heck, MD, Principal Investigator — Technical University of Munich; Christof Winter, MD PhD, Principal Investigator — Technical University of Munich
Locations (1):
- Technical University of Munich, Klinikum rechts der Isar, Department of Urology and Institute of Clinical Chemistry, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seitz AK, Thoene S, Bietenbeck A, Nawroth R, Tauber R, Thalgott M, Schmid S, Secci R, Retz M, Gschwend JE, Ruland J, Winter C, Heck MM. AR-V7 in Peripheral Whole Blood of Patients with Castration-resistant Prostate Cancer: Association with Treatment-specific Outcome Under Abiraterone and Enzalutamide. Eur Urol. 2017 Nov;72(5):828-834. doi: 10.1016/j.eururo.2017.07.024. Epub 2017 Aug 14. PMID 28818355